CLINICAL TRIAL: NCT01995825
Title: Evaluation of Bioequivalence of Lamotrigine Tablets in Epileptic Patients
Brief Title: Lamotrigine Bioequivalence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, James E Polli, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HP-00048923; HHSF223201010144A (Other Grant/Funding Number: HHS)
Record Dates: First submitted 2013-01-26; First posted 2013-11-27 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Epilepsy
Keywords: bioequivalence; lamotrigine; epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brand lamotrigine then Generic lamotrigine (Experimental): Crossover trial. Each arm will receive Brand lamotrigine tablet for two periods and Generic lamotrigine for two periods.
  Interventions: Drug: Brand lamotrigine; Drug: Generic lamotrigine
- Generic lamotrigine then Brand lamotrigine (Experimental): Crossover trial. Each arm will receive Generic lamotrigine tablet for two periods and Brand lamotrigine for two periods.
  Interventions: Drug: Brand lamotrigine; Drug: Generic lamotrigine

INTERVENTIONS:
Drug: Brand lamotrigine — Brand lamotrigine tablet 100mg tablets (1-3 either once or twice a day) for two weeks
Drug: Generic lamotrigine — Generic lamotrigine tablet 100mg tablets (1-3 either once or twice a day) for two weeks

SUMMARY:
In this study, brand name lamotrigine (LAMICTAL) and generic lamotrigine will be compared in patients with epilepsy. Both the brand name and generic lamotrigine are approved by the Food and Drug Administration (FDA) and are commonly used to treat epilepsy. Some physicians and patients with epilepsy have believed that brand and generic lamotrigine have had clinically significant differences in efficacy and tolerability. The brand name and generic tablets have been shown to be the same when blood levels were measured in healthy volunteers without epilepsy, but these drugs have not yet been compared in patients with epilepsy. This study will do this comparison, by switching patients between brand and generic in a very structured manner, and seeing if the drugs are the same, primarily in terms of blood levels. Other comparisons will also be made secondarily, looking for any differences in adverse effects and seizure control.

DETAILED DESCRIPTION:
As is commonly done in a bioequivalence study, the null hypothesis is that the generic (i.e. test) is bioINequivalent to the brand name (i.e. reference). Hence, the alternative hypothesis is that the generic is bioequivalent to the brand name.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent.
* Subject is male or female between 18 and 65 years of age inclusive.
* Subject has a diagnosis of epilepsy with simple partial seizures and/or complex partial seizures, with or without secondary generalization or primary generalized seizures.
* Subject has had a history of at least one seizure and/or AED related adverse event with AED changes; or had at least one seizure and/or AED related adverse event over the 12 months prior to Visit 1.
* Subject has been maintained on a stable dose regimen of anti-epileptic drugs (AEDs), including lamotrigine at 200mg, 400mg, or 600mg total daily dosage divided BID for at least 28 days prior to Visit 1. Additionally, subject must be taking lamotrigine for 8 weeks prior to Visit 1.
* Subject is willing to be switched between brand and generic lamotrigine.
* Subject is an acceptable candidate for venipuncture.
* Subject is willing to stop all OTC medications for 24 hours prior to and during 12 hour study visits.

Exclusion Criteria:

* Subject is currently participating or has participated within the last 2 months in any trial of an investigational drug or experimental device.
* Subject has a history of status epilepticus within the 12 month period prior to Visit 1.
* Subject has any medical condition, which in the opinion of the investigator, could jeopardize the subject's health or would compromise the subject's ability to participate in the trial.
* Subject has any psychiatric condition, which in the opinion of the investigator, could jeopardize the subject's health or would compromise the subject's ability to participate in this trial or confound the interpretation of the trial data.
* Subject has known hypersensitivity to lamotrigine.
* Subject has a medical condition that impacts drug absorption (e.g. gastric bypass surgery), including routine use (i.e. daily or weekly) use of acid blockers, antacids, anti-diarrhea, stimulants, appetite suppressants, or anti nausea medication or other drugs that modulate GI function.
* Subject has any history of alcohol or drug abuse within the previous two years.
* Subject has acute or subacutely progressive CNS disease.
* Subject has moderate or severe liver impairment as assessed by alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin levels ≥5 times the upper limit of normal (ULN).
* Subject has moderate or severe renal impairment as assessed by creatinine clearance lower than 50mL/min, using the Cockcroft-Gault formula.
* Female subjects of childbearing potential will not be eligible to participate who are unwilling or unable to use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: condom with spermicide, diaphragm with spermicide, IUD without progesterone, vaginal spermicidal suppository, surgical sterilization of their partner(s) or abstinence.
* Female subject is pregnant or nursing.
* Female subject is using hormonal contraceptive precautions including progesterone-coated IUD.
* Subjects is using hormonal replacement therapy.
* Subject is unwilling or unable to maintain their approximate daily smoking use during the study.
* Subject is using rifampin or other non-AED that strongly modulates lamotrigine levels.
* In addition to lamotrigine and/or vagus nerve stimulation and/or intermittent benzodiazepine use (e.g. lorazepam, diazepam, clonazepam), subject is taking more than two concomitant AEDs.
* Subject is not willing or able to be adherent to study protocol (e.g. dosing of lamotrigine and any interacting comedication).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

REFERENCES:
- [Background] Andermann F, Duh MS, Gosselin A, Paradis PE. Compulsory generic switching of antiepileptic drugs: high switchback rates to branded compounds compared with other drug classes. Epilepsia. 2007 Mar;48(3):464-9. doi: 10.1111/j.1528-1167.2007.01007.x. PMID 17346246

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brand Lamotrigine Then Generic Lamotrigine | Generic Lamotrigine Then Brand Lamotrigine
Started | 18 | 17
Completed | 17 | 17
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brand Lamotrigine Then Generic Lamotrigine | Generic Lamotrigine Then Brand Lamotrigine | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: pharmacokinetic exposure (ng*hr/ml)
Time Frame: 0-12hr
Measure: Mean (Standard Error); unit: ng*hr/ml
Groups:
- Brand Lamotrigine: Brand lamotrigine tablet100mg tablets (1-3 either once or twice a day) for two weeks
- Generic Lamotrigine: Generic lamotrigine tablet100mg tablets (1-3 either once or twice a day) for two weeks
Arm/Group | Brand Lamotrigine | Generic Lamotrigine
Number analyzed (Participants) | 34 | 34
ng*hr/ml | 101346 (6314) | 101393 (6421)

2. Primary Outcome: Cmax
Description: highest concentration over the time duration 0-12hr (ng/ml)
Time Frame: 0-12hr
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Brand Lamotrigine | Generic Lamotrigine
Number analyzed (Participants) | 34 | 34
ng/ml | 10670 (657) | 10697 (717)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Brand Lamotrigine | Generic Lamotrigine
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 7/35 | 6/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brand Lamotrigine (N=35) | Generic Lamotrigine (N=35)
headache (Nervous system disorders) | 4 (8) | 4 (5)
dizziness (Nervous system disorders) | 2 (3) | 2 (4)
nausea (General disorders) | 2 (2) | 1 (2)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
blurred vision (Ear and labyrinth disorders) | 1 (1) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No